CLINICAL TRIAL: NCT06139679
Title: Improvement In Left Ventricular Diameter After Closure Of Atrial Septal Defect With Fenestrated Patch: A Cross-sectional Study
Brief Title: Improvement In Left Ventricular Diameter After Closure Of ASD With Fenestrated Patch: A Cross-sectional Study
Status: Completed | Type: Observational
Sponsor: Dr. Soetomo General Hospital (Other Government)
Responsible Party: Principal Investigator, dr. Heroe Soebroto, Sp.B, Sp.BTKV, Subsp.JPK(K), MD, Dr. Soetomo General Hospital
Other Study IDs: 1148/110/3/XII/2021
Record Dates: First submitted 2023-11-02; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Atrial Septal Defect
Keywords: Left Ventricle Diameter; Atrial septal defect closure; Fenestrated patch
MeSH Terms: conditions — Heart Septal Defects, Atrial

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fenestrated: Patients with ASD who underwent surgical closure of ASD with fenestrated patch
  Interventions: Procedure: ASD closure with fenestrated/non-fenestrated patch
- Non-fenestrated: Patients with ASD who underwent surgical closure of ASD with non-fenestrated patch
  Interventions: Procedure: ASD closure with fenestrated/non-fenestrated patch

INTERVENTIONS:
Procedure: ASD closure with fenestrated/non-fenestrated patch — A PTFE patch is used to surgically close the interatrial defect. If closure with fenestrated patch is deemed necessary, a small opening is created on the patch

SUMMARY:
Introduction: The presence of pulmonary hypertension (PH) in atrial septal defect (ASD) poses a clinical challenge on whether or not to close the defect. Closing the defect increases the risk of low cardiac output syndrome (LCOS), while leaving the defect open may eventually lead to irreparable shunt reversal, hypoxemia, and death. The implementation of a fenestrated patch may halt LCOS while adding volume to the left heart.

Methods: this is an analytical observational study involving patients with ostium secundum defect with PH who were operated on in Dr. Soetomo Hospital between January 2017 and October 2021. The aim of this study is to evaluate the improvement in left ventricular size during both systole and diastole.

DETAILED DESCRIPTION:
Atrial septal defect (ASD) is one of the most common congenital heart diseases. It is typically characterized by a left-to-right shunt which results in volume overload of the right ventricle and overcirculation of the pulmonary vascularization (le Gloan et al., 2018). This may further result in arrhythmia, right ventricular dysfunction, and pulmonary hypertension (PH). Pulmonary hypertension is caused by endothelial dysfunction, remodelling of the pulmonary vascularization, which increases pulmonary vascular resistance, and eventually causes shunt reversal into right-to-left (Eisenmenger's syndrome). At this point, closure of the defect is contraindicated.

Small LV, although less extensively studied than dilated LV, also implies impaired LV function. Small LV means less tolerance to volume overload, which in turn impairs cardiac output and presents higher risk of heart failure and mortality (Saito et al., 2021).

ASD closure in cases with severe pulmonary hypertension (PH) presents a clinical challenge. Complete closure may cause pulmonary hypertensive crisis and low cardiac output syndrome; however, if left untreated, the disease progresses, the pulmonary vascular resistance increases, which may also lead to Eisenmenger's syndrome and shunt reversal. Today, this condition is treated with fenestrated closure, either with patch or fenestrated septal occluder. The fenestration is hypothesized to provide protective effect against pulmonary hypertensive crisis because it allows blood to flow from right to left heart. The added volume into the left heart is then, hypothesized, to provide volume training for the left heart, mainly in the case of small LV. Therefore, this study aims to evaluate the effect of fenestrated closure compared to non- fenestrated closure to the left ventricular size at systole and diastole.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ASD secundum and pulmonary hypertension with complete preoperative and postoperative echocardiography (LVIDd and LVIDs) data
* Patients with ASD secundum and pulmonary hypertension with complete preoperative but incomplete postoperative echocardiography (LVIDd and LVIDs) data, but willing to present upon invitation to complete missing postoperative data

Exclusion Criteria:

* Patients with ASD secundum and pulmonary hypertension who are unwilling to participate in the study, or in a condition that prevents the patient to present for echocardiographic evaluation
* Patients with incomplete medical records

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with ASD secundum with pulmonary hypertension of all age groups who underwent surgical closure of ASD in Dr. Soetomo General Academic Hospital within January 2017 - October 2021
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Improvement in left ventricular diameter during systole and diastole | January 2017 - October 2021
  The change in left ventricular diameter during both systole and diastole is measured preoperatively and postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Heroe Soebroto, Principal Investigator — Department of Thoracic, Cardiac, and Vascular Surgery, Dr. Soetomo General Hospital, Surabaya, Indonesia
Locations (1):
- Dr. Soetomo General Academic Hospital, Surabaya, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided